CLINICAL TRIAL: NCT06169358
Title: Screening Patients With Fabry Disease in Patients With Hypertrophic Cardiomyopathy or Left Ventricular Hypertrophy
Acronym: SEARCH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Other Study IDs: KYLL-202306-100-3
Record Dates: First submitted 2023-12-05; First posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-10

CONDITIONS: Hypertrophic Cardiomyopathy; Left Ventricular Hypertrophy; Fabry Disease
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Hypertrophy, Left Ventricular; Fabry Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples were collected for NT-proBNP values, routine blood tests (white blood cell count, hemoglobin, red blood cell count, platelet count, hematocrit), blood biochemistry (alanine aminotransferase, glutamine aminotransferase, urea nitrogen, creatinine, albumin, lipids, electrolytes, etc.), inflammatory markers (C-reactive protein, calcitonin), thyroid function (FT3, FT4, TSH, etc.), and markers of myocardial injury (troponin I, troponin T, creatine kinase isozymes, D-dimer, etc.), as well as genetic testing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study was to understand the epidemiological status of Fabry in patients with hypertrophic cardiomyopathy or left ventricular hypertrophy through multi-center early identification of high-risk patients in cardiology according to high-risk profiles, supplemented by DBS (dried blood disc) screening tools, and to explore the screening and diagnosis methods of patients with Fabry disease in cardiology, so as to promote the early identification, diagnosis and treatment of Fabry in cardiology.

ELIGIBILITY:
Inclusion Criteria:

* Meet diagnostic criteria for hypertrophic cardiomyopathy (HCM) in adults (age ≥ 18 years):Imaging of one or more left ventricular segments reveals a maximum end-diastolic ventricular wall thickness of ≥15 mm or end-diastolic ventricular septal thickness or posterior left ventricular wall thickness of ≥13 mm on either cardiac imaging at rest.

Exclusion Criteria:

* 1. Identification of hypertrophic cardiomyopathy caused by mutations in pathogenic genes; 2. Identify the cause of left ventricular hypertrophy (LVH); 3. Aortic valve or mitral valve lesions that can cause hemodynamic changes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Clinical case collection of patients with hypertrophic cardiomyopathy or left ventricular hypertrophy
Sampling Method: Non-Probability Sample
Enrollment: 627 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
diagnosis of Fabry disease | 1 year
  Clinicians can identify high-risk patients in cardiology at an early stage according to the high-risk profile developed in this study, supplemented by the DBS (dried blood disc) screening tool, and diagnose and treat Fabry disease as early as possible through the established screening pathway for high-risk patients with Fabry disease in cardiology.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoping Ji, Study Chair — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Jinan, China